CLINICAL TRIAL: NCT01677494
Title: To Assess the 12-month Prognostic Significance of Left Ventricular Collagen Markers in Patients With Heart Failure and Preserved Ejection Fraction.
Brief Title: Collagen Markers in Heart Failure and Preserved Ejection Fraction
Acronym: COLLAG4
Status: Terminated | Type: Observational
Why Stopped: lack of recruitment
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2010/068/HP
Record Dates: First submitted 2010-12-02; First posted 2012-09-03 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-09

CONDITIONS: Left-sided Congestive Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Proteomics
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- heart failure with preserved ejection fraction: - Inclusion Elevated BNP EF > 50%

SUMMARY:
Assessment of cardiac fibrosis by echocardiography (Speckle tracking), IRM (late-enhancement imaging), biology (markers of collagen turn-over) and proteomics

DETAILED DESCRIPTION:
Heart failure (HF) is a growing public health problem. While HF with deteriorated ejection fraction has faced numbers of (non) pharmacological advances, HF with preserved ejection fraction, which represents half of admission has today no efficient treatment.

Fibrosis is found in heart of patients with HF and preserved ejection fraction, is reponsible for stiff heart and has link to the transition to compensated/decompaseted HF and death.

The purpose of this work is to characterise myocardial fibrosis by any means to change the prognosis of patients with HF and preserved ejection fraction

Main purpose:

Assessment of cardiac fibrosis by echocardiography (Speckle tracking), IRM (late-enhancement imaging), biology (markers of collagen turn-over) and proteomics

* Patients selection

  1. - Inclusion Criteria: Male or female > 18 and < 85 years of age. Recent HF decompensation (framingham criteria, ejection fraction > 50% with 72 hours after admission and BNP > 100 ng/L or NT-proBNP > 300 ng/L), signed inform consent.
  2. - exclusion criteria: hypertrophic cardiomyopathy, restrictive cardiomyopathy, constrictive pericarditis, significant respiratory disease, pulmonary hypertension, core pulmonale, end-stage kidney disease, high cardiac output HF, isolated right ventricular dysfunction, pregnancy or child-bearing, biventricular pacing, No health insurance.
* Control group

  1. - inclusion criteria: Male or female > 18 and < 85 years of age. signed inform consent. Health insurance.
  2. - exclusion criteria: significant ischemic heart disease, significant valvular heart disease, pericarditis, pulmonary hypertension, hypertrophic cardiomyopathy, restrictive cardiomyopathy, constrictive pericarditis, significant respiratory disease, pulmonary hypertension, core pulmonale, end-stage kidney disease, high cardiac output HF, isolated right ventricular dysfunction, pregnancy or child-bearing, biventricular pacing, No health insurance.

ELIGIBILITY:
- inclusion Signs of heart failure Elevated BNP EF > 50% within 72 hours after admission

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: heart failure with preserved ejection fraction
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2010-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
death and admission for heart failure | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice Bauer, MD, PhD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen university hospital, Rouen, France